CLINICAL TRIAL: NCT04948463
Title: Early Versus Late Stopping of Antibiotics in Children With Cancer and High-risk Febrile Neutropenia
Acronym: ELSA-FN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 74690
Record Dates: First submitted 2021-06-18; First posted 2021-07-02 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-11

CONDITIONS: Febrile Neutropenia
Keywords: Febrile Neutropenia; Cancer; Haematopoietic Stem Cell Transplantation (HSCT)
MeSH Terms: conditions — Febrile Neutropenia; Neoplasms | interventions — Piperacillin; Tazobactam; Injections; Cefepime; Ceftazidime; Vancomycin; Amikacin; Ciprofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early Stopping (Experimental): Stopping empiric FN antibiotics after resolution of fever for 48 hours, irrespective of absolute neutrophil count (ANC)
  Interventions: Drug: Piperacillin and Tazobactam for Injection; Drug: Cefepime Injection; Drug: Ceftazidime Injection; Drug: Vancomycin Injection; Drug: Amikacin Injection; Drug: Ciprofloxacin
- Standard of care (Active Comparator): Continuing empiric FN antibiotics until resolution of fever for 48 hours and recovery of ANC as defined by the treating clinician but usually to ≥200-500/mm3
  Interventions: Drug: Piperacillin and Tazobactam for Injection; Drug: Cefepime Injection; Drug: Ceftazidime Injection; Drug: Vancomycin Injection; Drug: Amikacin Injection; Drug: Ciprofloxacin

INTERVENTIONS:
Drug: Piperacillin and Tazobactam for Injection — Given if patient has no known allergies, until ANC recovery at 100mg/kg (max 4g) 6 hourly.
  Arms: Standard of care
Drug: Cefepime Injection — Given if patient has non life-threatening hypersensitivity (preferred option), until ANC recovery at 50mg/kg (max 2g) 8 hourly.
  Arms: Standard of care
Drug: Ceftazidime Injection — If non life-threatening hypersensitivity (second option), given until ANC recovery at 50mg/kg (max 2g) 8 hourly
  Arms: Standard of care
Drug: Vancomycin Injection — If life-threatening hypersensitivity given with ciprofloxacin, given until ANC recovery at 15mg/kg (max 500mg) 6 hourly
  Arms: Standard of care
Drug: Amikacin Injection — Given until ANC recovery at 18-22.5mg/kg (max 1.5g) daily in combination with other antibiotic/s.
  Arms: Standard of care
Drug: Ciprofloxacin — If life-threatening hypersensitivity given with vancomycin, given until ANC recovery at 10 mg/kg (max 400 mg) 12 hourly
  Arms: Standard of care
Drug: Piperacillin and Tazobactam for Injection — Given if patient has no known allergies at 100mg/kg (max 4g) 6 hourly, stopping 48 hours post-fever resolution.
  Arms: Early Stopping
Drug: Cefepime Injection — If non life-threatening hypersensitivity (preferred option) at 50mg/kg (max 2g) 8 hourly, stopping 48 hours post-fever resolution
  Arms: Early Stopping
Drug: Ceftazidime Injection — If non life-threatening hypersensitivity (second option) at 50mg/kg (max 2g) 8 hourly, stopping 48 hours post-fever resolution
  Arms: Early Stopping
Drug: Vancomycin Injection — If life-threatening hypersensitivity given with ciprofloxacin at 15mg/kg (max 500mg) 6 hourly, stopping 48 hours post-fever resolution
  Arms: Early Stopping
Drug: Amikacin Injection — At 18-22.5mg/kg (max 1.5g) daily in combination with other antibiotic/s, stopping 48 hours post-fever resolution
  Arms: Early Stopping
Drug: Ciprofloxacin — If life-threatening hypersensitivity given with vancomycin at 10 mg/kg (max 400 mg) 12 hourly, stopping 48 hours post-fever resolution
  Arms: Early Stopping

SUMMARY:
This randomised controlled trial will determine the non-inferiority of stopping empiric antibiotics prior to absolute neutrophil count (ANC) recovery (Early Stopping) versus stopping antibiotics upon ANC recovery (Standard of Care/ Late Stopping) , in children with cancer and high-risk febrile neutropenia (FN).

DETAILED DESCRIPTION:
Febrile neutropenia (FN) is a common complication of childhood cancer treatment and a leading cause of hospital admission and antibiotic exposure. Management typically involves broad-spectrum antibiotics until resolution of fever and absolute neutrophil count (ANC) recovery >500 cells/mm3. However, despite the frequency with which FN occurs, evidence to guide duration of antibiotics is limited to observational studies and small randomised controlled trials.Current international clinical guidelines provide conflicting recommendations on when to cease empiric antibiotics for FN. Early cessation of antibiotics in FN may translate to reduced antibiotic exposure and limit potential harms including drug side-effects, antimicrobial resistance, Clostridioides difficile infection and microbiome disruption. This randomised controlled trial will use a composite endpoint of fever recurrence, physiological instability, new bacteremia, intensive care admission and death to determine the non-inferiority of stopping antibiotics prior to ANC recovery compared with standard of care (SOC), in children with cancer and high-risk FN. Adopting a health informatics approach, patient identification, consent, randomisation and reporting of outcomes will be embedded within the electronic medical record (EMR). Children with high-risk FN who have been afebrile and clinically stable for at least 48 hours will be randomised to cease antibiotics or continue SOC. Data on primary outcomes, antibiotic duration, length of stay, C. difficile infection and antimicrobial resistance will be automatically collected by the EMR. This is the first study of its kind in children with high-risk FN and adopts a novel embedded trial design. Results will inform optimal antibiotic duration in FN, potentially reducing unnecessary antibiotic exposure.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of

   * Acute myeloid leukemia (AML) or acute lymphoblastic leukaemia (ALL) in dose-intensive phases of induction/re-induction, intensification or consolidation or
   * ALL or acute lymphoblastic lymphoma patients on a TOT17 protocol or
   * Any disease within 100 days of allogeneic or autologous HSCT
2. Neutropenia (<500 cells/mm3)
3. Afebrile (temperature <38.0°C) period for at least 48 hours and no more than 96 hours after at least one temperature measured by axillary or tympanic thermometer (≥38.0°C)
4. Commenced on empiric FN antibiotics (any of piperacillin-tazobactam, cefepime, ceftazidime or vancomycin and ciprofloxacin)

Exclusion Criteria:

1. Prolonged febrile neutropenia (documented daily temperature ≥38.0°C for ≥5 days)
2. Documented positive blood culture since onset of FN episode and prior to randomisation
3. Documented other infection (microbiologically or clinically documented) requiring antibiotic treatment since onset of FN episode and prior to randomisation
4. Admitted to the ICU at the time of randomisation
5. Clinical instability (One or more conscious state, respiratory rate, blood pressure, heart rate or oxygen saturations in MET criteria OR two or more respiratory rate, blood pressure, heart rate or oxygen saturations simultaneously (+/- 4 hrs) in the clinical review criteria in 48 hours prior to randomisation)
6. Within 28 days of last randomisation

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 55 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2025-12-17 (Actual); Study Completion 2025-12-17 (Actual)

PRIMARY OUTCOMES:
Unfavourable clinical course occurring during the same period of severe neutropenia | During the same episode of neutropenia, up to 28 days post-enrolment.
  Incidence of unfavourable clinical course, defined as any of the following: recurrence of fever, clinical instability (see below definition), admission to the intensive care unit, new positive blood culture collected after randomisation, or death

SECONDARY OUTCOMES:
Fever recurrence | Up to 28 days post-enrolment
  Incidence of fever recurrence (temperature ≥38 degrees Celsius)
Clinical instability | Up to 28 days post-enrolment
  Incidence of clinical instability defined as; one or more vital signs (conscious state, respiratory rate, blood pressure, heart rate, oxygen saturation) meeting mandatory emergency (MET) call criteria OR two or more vital signs simultaneously (within 4 hours of each other) meeting clinical review criteria.
Admission to intensive care unit (ICU) | Up to 28 days post-enrolment
  Incidence of admission to intensive care unit (all cause)
New positive blood culture | Up to 28 days post-enrolment
  Incidence of positive blood culture
28 day all-cause and infection-related mortality | Up to 28 days post-enrolment
  Incidence of all-cause and infection-related mortality, as defined post-mortem
Duration of neutropenia | During the same episode of neutropenia or up to 28 days post-enrolment
  Mean days of neutropenia defined as ANC <500 cells/mm3
Clinician confidence and acceptability | Up to 28 days post-enrolment
  Measured by number of patients for which randomisation is overridden in the Early Stopping arm and the recorded reason
Total antibiotic duration | Up to 28 days post-enrolment
  Mean number of days antibiotics are administered
Length of hospital stay | Up to 28 days post-enrolment, or until discharge from hospital (whichever is the later)
  Mean number of days admitted to the study site hospital ward
Readmission to hospital | Up to 28 days post-enrolment
  Incidence of unplanned admission to the study site hospital
Development of C. difficile infection | Up to 28 days post-enrolment
  Incidence of C. difficile infection detected in unformed stool
Development of an antibiotic resistant infection or colonisation | Up to 28 days post-enrolment
  Incidence of antibiotic resistant infection or colonisation including Methicillin-resistant Staphylococcus aureus (MRSA), extended spectrum beta-lactamases (ESBL)-producing enterobacterales, carbapenem-resistant enterobacteriaceae (CRE), Vancomycin-resistant Enterococcus (VRE)
Patient/parent/caregiver confidence | Within 48 hours of having informed consent discussion with the study team
  Number of patients that consent to study as proportion of patients eligible
Patient/parent/caregiver acceptability | Within 48-96 hours post assignment to intervention arm
  Number of patients for which randomisation is overridden in the Early Stopping arm due to withdrawn consent

CONTACTS AND LOCATIONS:
Overall Officials: Gabrielle Haeusler, Principal Investigator — Murdoch Childrens Research Institute
Locations (1):
- Royal Children's Hospital, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
Beginning 6 months following analysis and publication of the primary outcome, data will be made available long-term for use by future researchers from a recognised research institution whose proposed use of the data has been ethically reviewed and approved by the Murdoch Children's Research Institute's (MCRI's) independent data use review committee (not including trial sponsor-investigator) and who accept MCRI's conditions, under a collaborator agreement, for accessing all of the available participant data collected during the trial (after full deidentification).
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: 6 months following analysis and publication of the primary outcome
Access Criteria: Requests for access to previously published anonymised datasets by the scientific community will be reviewed and determined by an independent committee within the MCRI and in accordance with institute policy.